CLINICAL TRIAL: NCT01420497
Title: Systemic Effects of Epidural Methylprednisolone Injection on Glucose Tolerance in Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, zufferey Pascal, md, Centre Hospitalier Universitaire Vaudois
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: gylperi
Record Dates: First submitted 2011-08-18; First posted 2011-08-19 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-08

CONDITIONS: Diabetes; Healthy
Keywords: methylprednisolone; intra articular infiltration; glycemia; epidural infiltration; diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- methylprednisolone,infiltration (Active Comparator)
  Interventions: Drug: intra-articular infiltration
- epidural injection (Active Comparator)
  Interventions: Drug: epidural infiltration

INTERVENTIONS:
Drug: intra-articular infiltration — intra articular infiltration
  Arms: methylprednisolone,infiltration
Drug: epidural infiltration — epidural infiltration
  Arms: epidural injection

SUMMARY:
Several studies have shown that in diabetic patients, the glycemic profile was disturbed after intra-articular injection of corticosteroids. Little is known about the impact of epidural injection in such patients. The goal of this study was double, at first comparing the glycaemic profile in diabetic patients after a unique injection of 80 mg of acetate methylprednisolone either intra-articular or epidural, secondly to compare the amount of systemic diffusion of the drug the after both procedures.

ELIGIBILITY:
Inclusion Criteria:

* diabetes stable for more than ten days
* no contraindication for steroids
* lumbar stenosis
* articular pain

Exclusion Criteria:

* unstable diabetes
* renal insufficiency

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-08; Primary Completion 2008-09 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
glycemic values, | day 0 to day 15

SECONDARY OUTCOMES:
urinary excretion rate | day 0 to day 15

CONTACTS AND LOCATIONS:
Locations (1):
- CHUV, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Zufferey P, Bulliard C, Gremion G, Saugy M, So A. Systemic effects of epidural methylprednisolone injection on glucose tolerance in diabetic patients. BMC Res Notes. 2011 Dec 21;4:552. doi: 10.1186/1756-0500-4-552. PMID 22185681